CLINICAL TRIAL: NCT03653182
Title: The Relation Between Constitutional Types and Indices of Tongue, Pulse,and Ausculative Diagnosis
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: Committee on Chinese Medicine and Pharmacy (Other Government)
Responsible Party: Sponsor
Other Study IDs: DMR99-IRB-271
Record Dates: First submitted 2018-07-09; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Non-disease State
MeSH Terms: interventions — Pulse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- normal: A normal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Qi deficiency: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Damp heat: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Yang deficiency: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Yin deficiency: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Phlagm: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Blood stasis: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Qi stagnation: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound
- Special: One of an abnormal constitution condition in TCM.
  Interventions: Diagnostic Test: Pulse, tongue image, and voice sound

INTERVENTIONS:
Diagnostic Test: Pulse, tongue image, and voice sound — They are four diagnosis methods of TCM

SUMMARY:
This study aims to evaluate indices of tongue diagnosis, ausculative diagnosis, and pulse diagnosis in the determination of institutions.

DETAILED DESCRIPTION:
Constitution differentiation is important for the prescription of Chinese medicines. In previous studies, researchers usually used constitutional questionnaires to determine constitutions.However, the importance of tongue diagnosis and pulse diagnosis remained unclear. The specific aim of this study is to evaluation indices of tongue diagnosis, auscultative diagnosis, and pulse diagnosis in the determination of constitutions. Meeting of specialists will determine the characteristics for each constitution first. This study plans to recruit 200 volunteers and determine their constitutions by constitutional questionnaires. Tongue manifestations and pulse pressure waveforms will be taken at the same time by standardized instruments. Relations between the indices and each constitution will be determined by multiple linear regression and logistic regression analysis. Then the percentage of importance of a specific index in a specific constitutional type could be determine.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers without aged older than 20 years old

Exclusion Criteria:

* Pregnant
* taking any medicine currently
* suffering for acute disease currently

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aged older than 20 years old
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2010-12-15 (Actual); Primary Completion 2011-12-14 (Actual); Study Completion 2011-12-14 (Actual)

PRIMARY OUTCOMES:
Tongue image | The photograph will be taken only at the first day the subject has been recruited
  A photograph of tongue will be taken and the RGB color values of the tongue will be analyzed using Photoshop software

SECONDARY OUTCOMES:
Acoustic sound | The voice waves will be taken only once at the first day the subject has been recruited
  Voice wave analysis of an one-second /a/ sound (in only one time point)
Pulse image | The pulse waveforms will be recorded at the first day the subject has been recruited
  Time-domained pulse waveform of the radial artery will be recorded for about 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- CMUH, Taichung, Taiwan